CLINICAL TRIAL: NCT00433511
Title: A Double-Blind Phase III Trial of Doxorubicin and Cyclophosphamide Followed by Paclitaxel With Bevacizumab or Placebo in Patients With Lymph Node Positive and High Risk Lymph Node Negative Breast Cancer
Brief Title: Doxorubicin Hydrochloride, Cyclophosphamide, and Paclitaxel With or Without Bevacizumab in Treating Patients With Lymph Node-Positive or High-Risk, Lymph Node-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00561; NCI-2009-00561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000528955; E5103; ECOG-E5103; 07-963; E5103 (Other: ECOG-ACRIN Cancer Research Group); E5103 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Adenocarcinoma
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (chemotherapy, placebo) (Active Comparator): Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV over 20-30 minutes, and placebo IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel IV over 1 hour on days 1, 8, and 15 and placebo IV over 30-90 minutes on day 1. Treatment with paclitaxel and placebo repeats every 3 weeks for 4 courses.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo Administration; Other: Quality-of-Life Assessment
- Arm II (chemotherapy, bevacizumab) (Experimental): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm III (chemotherapy, bevacizumab monotherapy) (Experimental): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I and bevacizumab as in arm II. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm I and bevacizumab as in arm II. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses. Beginning 2 months later, patients then receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab alone repeats every 3 weeks for 10 courses.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm II (chemotherapy, bevacizumab); Arm III (chemotherapy, bevacizumab monotherapy)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo Administration — Given IV
  Arms: Arm I (chemotherapy, placebo)
Other: Quality-of-Life Assessment — Ancillary studies (closed as of 5/28/10)
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies doxorubicin hydrochloride, cyclophosphamide, and paclitaxel to see how well they work with or without bevacizumab in treating patients with cancer that has spread to the lymph nodes (lymph node-positive) or cancer that has not spread to the lymph nodes but is at high risk for returning (high-risk, lymph node-negative breast cancer). Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery and help prevent the tumor from returning. It is not yet known whether doxorubicin hydrochloride, cyclophosphamide, and paclitaxel are more effective with or without bevacizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the disease-free survival of patients (defined as invasive disease-free survival [IFDS]) with lymph node positive and high risk lymph node negative breast cancer randomized to treatment with either doxorubicin (doxorubicin hydrochloride)/cyclophosphamide plus placebo followed by paclitaxel (AC + placebo > T + placebo) or the same chemotherapy regimen plus bevacizumab.

SECONDARY OBJECTIVES:

I. To compare short-term (20-24 weeks) versus long-term (50-54 weeks) bevacizumab therapy.

II. To compare the overall survival. III. To evaluate toxicity. IV. To evaluate the association between outcomes in E5103 (disease-free survival, overall survival and toxicities) and genotype (derived from candidate single nucleotide polymorphisms and genome wide evaluations).

V. To compare the quality of life of breast cancer patients treated with AC/paclitaxel and bevacizumab or placebo, in terms of physical symptoms, physical functioning, psychological state and social functioning over an 18 month period.

VI. To determine the impact of theoretical biomarker information on patients' willingness to accept the toxicities of bevacizumab for the estimated potential benefit.

VII. To create a biospecimen repository including plasma, serum and CellSearch cassettes containing circulating tumor cells (CTC) for evaluating determinants of late relapse, including candidate biomarkers reflecting occult tumor burden (e.g., CTCs and plasma tumor deoxyribonucleic acid [DNA]) and host factors (e.g., estrogen, insulin-insulin-like growth factor [IGF] axis, inflammation, etc).

VIII. To create a biorepository of metastatic tumor samples in patients who have had a late relapse.

IX. To determine body mass index (BMI) and comorbidity burden in patients with operable breast cancer five or more years after diagnosis.

X. To determine whether there is a relationship between late relapse and BMI at diagnosis and at 5 years after diagnosis, and whether BMI-associated inflammatory and/or metabolic biomarkers are associated with early and late recurrence.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive doxorubicin hydrochloride intravenously (IV), cyclophosphamide IV over 20-30 minutes, and placebo IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel IV over 1 hour on days 1, 8, and 15 and placebo IV over 30-90 minutes on day 1. Treatment with paclitaxel and placebo repeats every 3 weeks for 4 courses.

ARM II: Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses.

ARM III: Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I and bevacizumab as in arm II. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm I and bevacizumab as in arm II. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses. Beginning 2 months later, patients then receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab alone repeats every 3 weeks for 10 courses.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the breast at significant risk of distant recurrence based on at least one of the following criteria:

  * For axillary lymph node positive disease:

    * Involvement of at least one sentinel or axillary lymph node on routine histologic examination; patients with negative sentinel nodes and negative axillary nodes or involvement only demonstrated by immunohistochemistry are not eligible unless they meet one of the other eligibility criteria below
    * NOTE: consider intramammary nodes as equivalent to axillary nodes for the purposes of eligibility and stratification
  * For axillary lymph node negative disease:

    * Estrogen receptor (ER) negative tumor >= 1 cm
    * ER+ tumor >= 5 cm regardless of recurrence score
    * ER+ tumor >= 1 cm but < 5 cm with a recurrence score >= 11 (patients enrolled in the TAILORx trial are eligible)
    * NOTE: axillary dissection is strongly encouraged in patients with lymph node involvement identified on sentinel node biopsy
* Patients must have completed definitive breast surgery including total mastectomy and axillary dissection (modified radical mastectomy), total mastectomy and sentinel node biopsy, breast conservation surgery and axillary dissection or breast conservation surgery and sentinel node biopsy

  * NOTE: breast conservation surgery includes lumpectomy, partial mastectomy, and excisional biopsy
* Margins of breast conservation surgery or mastectomy must be histologically free of invasive breast cancer and ductal carcinoma in situ (DCIS); patients with resection margins positive for lobular carcinoma in situ (LCIS) are eligible
* Time from last surgery for breast cancer (breast conservation surgery, mastectomy, sentinel node biopsy, axillary dissection or re-excision of breast conservation surgery margins) to planned treatment start date must be > 28 days and =< 84 days
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Within =< 8 weeks prior to randomization: Absolute neutrophil count >= 1,000/mm^3
* Within =< 8 weeks prior to randomization: Platelet count >= 100,000/mm^3
* Within =< 8 weeks prior to randomization: Total bilirubin =< 1.5 mg/dL
* Within =< 8 weeks prior to randomization: Aspartate aminotransferase (AST) =< 2 times upper limit of normal(ULN)
* Within =< 8 weeks prior to randomization: Serum creatinine =< 1.5 mg/dL
* Within =< 8 weeks prior to randomization: Urine protein:creatinine ratio < 1.0 or 24-hour protein
* Within =< 8 weeks prior to randomization: Partial thromboplastin time (PTT) =< 1.5 times ULN
* Within =< 8 weeks prior to randomization: Left ventricle ejection fraction (LVEF) >= institutional limits of normal by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
* Patients who have undergone breast conservation surgery must receive radiation; prior to randomization, the investigator must specify the planned radiation technique:

  * Whole breast radiation (WBRT) after chemotherapy
  * Accelerated partial breast radiation (APBI) after chemotherapy
  * Accelerated partial breast radiation (APBI) prior to chemotherapy
  * NOTE: if APBI was completed prior to study entry, day 1 of protocol therapy must be at least 4 weeks after the completion of APBI
* Post-mastectomy radiation therapy (RT) is required for all patients with a primary tumor of >= 5 cm or involvement of 4 or more lymph nodes; post-mastectomy RT may be administered at the investigator's discretion for all other mastectomy patients
* Patients with human epidermal growth factor receptor (HER)2 + (3+ by immunohistochemistry [IHC] or fluorescent in situ hybridization [FISH] ratio >= 2) breast cancer are not eligible
* Patients with synchronous bilateral breast cancer (diagnosed within one month) are eligible if the higher tumor, node, metastasis (TNM) stage tumor meets the eligibility criteria for this trial
* Patients must not have clinical evidence of inflammatory disease or fixed axillary nodes at diagnosis
* Patients must not have received prior cytotoxic chemotherapy or hormonal therapy for this breast cancer; prior treatment with an anthracycline, anthracenedione or taxane for any condition is not allowed

  * NOTE: prior use of tamoxifen for chemoprevention is allowed but must be discontinued at study entry; similarly, prior raloxifene use is allowed but must be discontinued at study entry
* Patients must not have had any major surgical procedure within 28 days of planned treatment start date

  * NOTE: non-operative biopsy or placement of a vascular access device is not considered a major surgery
* Patients may not have had placement of a vascular access device within 24 hours of planned day 1 of treatment
* Patients must not have clinically significant cardiovascular or cerebrovascular disease, including:

  * Any history of

    * Cerebrovascular disease including transient ischemic attack (TIA), stroke or subarachnoid hemorrhage
    * Ischemic bowel
  * Within the last 12 months

    * Myocardial infarction
    * Unstable angina
    * New York Heart Association (NYHA) class II or greater congestive heart failure
    * Grade II or greater peripheral vascular disease
    * Uncontrolled hypertension defined as systolic blood pressure (SBP) > 160 or diastolic blood pressure (DBP) > 90
    * Uncontrolled or clinically significant arrhythmia
    * NOTE: blood pressure must be obtained within =< 8 weeks prior to randomization
    * NOTE: patients with controlled atrial fibrillation are eligible
* Patients who require full-dose anticoagulation may enroll provided they meet the following criteria:

  * The patient must have an in-range international normalized ratio (INR) (usually between 2 and 3) on a stable dose of warfarin or be on stable dose of low molecular weight (LMW) heparin
  * The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. varices)
  * NOTE: prophylactic use of anticoagulants to maintain patency of a vascular access device is permitted
* Patients must not have a bleeding diathesis, hereditary or acquired bleeding disorder or coagulopathy
* Patients must not have a non-healing wound or fracture; patients with an abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization are not eligible
* Patients must not have hypersensitivity to paclitaxel or drugs using the vehicle Cremophor, Chinese hamster ovary cell products or other recombinant human antibodies
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood or urine test within 7 days prior to randomization to rule out pregnancy
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4994 (Actual)
Dates: Start 2007-11-02 (Actual); Primary Completion 2014-01-07 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D Miller, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (843):
- United States (841):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - California Cancer Associates for Research and Excellence (cCare), Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Eisenhower Army Medical Center, Fort Eisenhower, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Bloomington, Bloomington, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Research LLC, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - York Hospital, York Village, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Missouri Cancer Care PC - Saint Charles, Saint Charles, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - San Juan Regional Medical Center, San Juan, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Queens Hospital Center, Jamaica, New York
  - Garnet Health Medical Center, Middletown, New York
  - Mount Kisco Medical Group at Northern Westchester Hospital, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - The Dyson Center for Cancer Care, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Derived] Rosenberg SM, O'Neill A, Sepucha K, Miller KD, Dang CT, Northfelt DW, Sledge GW, Schneider BP, Partridge AH. Quality of Life Following Receipt of Adjuvant Chemotherapy With and Without Bevacizumab in Patients With Lymph Node-Positive and High-Risk Lymph Node-Negative Breast Cancer. JAMA Netw Open. 2022 Feb 1;5(2):e220254. doi: 10.1001/jamanetworkopen.2022.0254. PMID 35226083
- [Derived] Ip EH, Saldana S, Miller KD, Carlos RC, Gareen IF, Sparano JA, Graham N, Zhao F, Lee JW, O'Connell NS, Cella D, Peipert JD, Gray RJ, Wagner LI. Tolerability of bevacizumab and chemotherapy in a phase 3 clinical trial with human epidermal growth factor receptor 2-negative breast cancer: A trajectory analysis of adverse events. Cancer. 2021 Dec 15;127(24):4546-4556. doi: 10.1002/cncr.33992. Epub 2021 Nov 2. PMID 34726788
- [Derived] Sparano J, O'Neill A, Alpaugh K, Wolff AC, Northfelt DW, Dang CT, Sledge GW, Miller KD. Association of Circulating Tumor Cells With Late Recurrence of Estrogen Receptor-Positive Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1700-1706. doi: 10.1001/jamaoncol.2018.2574. PMID 30054636
- [Derived] Miller KD, O'Neill A, Gradishar W, Hobday TJ, Goldstein LJ, Mayer IA, Bloom S, Brufsky AM, Tevaarwerk AJ, Sparano JA, Le-Lindqwister NA, Hendricks CB, Northfelt DW, Dang CT, Sledge GW Jr. Double-Blind Phase III Trial of Adjuvant Chemotherapy With and Without Bevacizumab in Patients With Lymph Node-Positive and High-Risk Lymph Node-Negative Breast Cancer (E5103). J Clin Oncol. 2018 Sep 1;36(25):2621-2629. doi: 10.1200/JCO.2018.79.2028. Epub 2018 Jul 24. PMID 30040523
- [Derived] Partridge AH, Sepucha K, O'Neill A, Miller KD, Baker E, Dang CT, Northfelt DW, Sledge GW, Schneider BP. Does biomarker information impact breast cancer patients' preferences and physician recommendation for adjuvant chemotherapy? Breast Cancer Res Treat. 2017 Oct;165(3):545-553. doi: 10.1007/s10549-017-4338-x. Epub 2017 Jun 23. PMID 28646344
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual to Step 1 of E5103 was activated November 2, 2007 and closed February 28, 2011; 4994 patients were entered. Upon unblinding of Step 1 treatment assignment, only patients treated on Arm C during Step 1 who had not ended protocol treatment early were eligible to register to Step 2 (Arm D) and 1316 patients were enrolled to Step 2.
Groups:
- Arm A (Chemo + Placebo): Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV over 20-30 minutes, and placebo IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel IV over 1 hour on days 1, 8, and 15 and placebo IV over 30-90 minutes on day 1. Treatment with paclitaxel and placebo repeats every 3 weeks for 4 courses.
- Arm B (Chemo + Bevacizumab): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm A and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm A and bevacizumab IV over 30-90 minutes on day 1. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses.
- Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm A and bevacizumab as in arm B. Treatment repeats every 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm A and bevacizumab as in arm B. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses. Within the following 2 months, patients then receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab alone repeats every 3 weeks for 10 courses. The monotherapy of bevacizumab is considered as arm D in this study.
Period: Step 1
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy)
Started | 1000 | 1986 | 2008
Patients Who Received Treatment | 972 | 1922 | 1942
Patients in Genetic Ancestry Analysis | 575 | 1126 | 1158
Completed | 864 | 1601 | 1618
Not Completed | 136 | 385 | 390
Not completed — Adverse Event | 50 | 157 | 153
Not completed — Withdrawal by Subject | 45 | 143 | 154
Not completed — Death | 3 | 1 | 1
Not completed — Physician Decision | 1 | 4 | 3
Not completed — Never started protocol therapy | 28 | 64 | 66
Not completed — Alternative therapy | 2 | 1 | 3
Not completed — Disease progression, relapse | 5 | 3 | 3
Not completed — Other complicating disease | 2 | 6 | 3
Not completed — Non-breast cancer surgery/wound issues | 0 | 4 | 1
Not completed — Suspected recurrence | 0 | 1 | 0
Not completed — Insurance/drug distribution issues | 0 | 1 | 2
Not completed — Patient moved | 0 | 0 | 1
Period: Step 2 (Arm D)
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy)
Started | 0 (Only Arm C patients at Step 1 who did not end protocol therapy early were eligible for Step 2, Arm D) | 0 (Only Arm C patients at Step 1 who did not end protocol therapy early were eligible for Step 2, Arm D) | 1316 (Only Arm C patients at Step 1 who did not end protocol therapy early were eligible for Step 2, Arm D)
Patients Who Received Treatment | 0 | 0 | 1168
Completed | 0 | 0 | 825
Not Completed | 0 | 0 | 491
Not completed — Adverse Event | 0 | 0 | 135
Not completed — Withdrawal by Subject | 0 | 0 | 181
Not completed — Never started protocol therapy | 0 | 0 | 148
Not completed — Physician Decision | 0 | 0 | 9
Not completed — Disease progression, relapse | 0 | 0 | 7
Not completed — Other complicating disease | 0 | 0 | 3
Not completed — Non-breast cancer surgery/wound issues | 0 | 0 | 2
Not completed — Suspected recurrence | 0 | 0 | 1
Not completed — Insurance/drug distribution issues | 0 | 0 | 4
Not completed — Unknown (Missing off treatment form) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm A and bevacizumab as in arm B. Treatment repeats every 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm A and bevacizumab as in arm B. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses. Beginning 2 months later, patients then receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab alone repeats every 3 weeks for 10 courses. The monotherapy of bevacizumab is considered as arm D in this study.
- Total: Total of all reporting groups
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy) | Total
Number analyzed (Participants) | 1000 | 1986 | 2008 | 4994
Age, Continuous [Median (Full Range); unit: years] | 51.8 [25.4 to 77.7] | 51.7 [21.2 to 85.0] | 51.6 [21.5 to 82.5] | 51.7 [21.2 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 995 | 1976 | 2000 | 4971
  Male | 5 | 10 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 136 | 160 | 366
  Not Hispanic or Latino | 891 | 1757 | 1752 | 4400
  Unknown or Not Reported | 39 | 93 | 96 | 228

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-free Survival (IDFS) Rate at 5 Years
Description: Invasive disease-free survival (IDFS) was defined as time from from date of randomization to first treatment failure (invasive ipsilateral, local/regional, or distant recurrence, invasive contralateral breast cancer, invasive non-breast second primary malignancy or death from any cause, whichever occurred first). Cases with incomplete follow-up, without documented IDFS event including those who developed squamous or basal cell skin cancers or insitu carcinomas of any site as their only event were censored at the date of last disease evaluation.
Time Frame: Assessed at 5 years
Population: All randomized patients at Step 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy)
Number analyzed (Participants) | 1000 | 1986 | 2008
proportion of participants | 0.77 [0.71 to 0.81] | 0.76 [0.72 to 0.80] | 0.80 [0.77 to 0.83]
Statistical Analysis 1: Comparison: Arm A (Chemo + Placebo) vs Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy); The primary objective of this trial was to determine whether the addition of bevacizumab improved IDFS. A two-step hierarchical approach was used. In the 1st step, Arm C was to be compared to Arm A. If Arm C significantly improved IDFS relative to Arm A, then in the 2nd step, a comparison of Arm B to Arm A was to be performed. If the treatment in both Arm C and Arm B significantly improved IDFS relative to Arm A, then a comparison of Arm C to Arm B was to be performed with respect to IDFS; Test type: Superiority; p = 0.17, Regression, Cox — Two-sided; based on stratified test using stratification factors at randomization; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.06] — Hazard ratio: Arm C/Arm A

2. Secondary Outcome: 5-year Overall Survival (OS)
Description: Overall survival (OS) was defined as time from date of randomization to death from any cause, otherwise cases were censored at date last known to be alive.
Time Frame: Assessed at 5 years
Population: All randomized patients at Step 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy)
Number analyzed (Participants) | 1000 | 1986 | 2008
proportion of participants | 0.90 [0.87 to 0.92] | 0.86 [0.83 to 0.88] | 0.90 [0.88 to 0.92]
Statistical Analysis 1: Comparison: Arm A (Chemo + Placebo) vs Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy); Test type: Superiority; p = 0.41, Regression, Cox — Two-sided; based on stratified test using stratification factors at randomization; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.68 to 1.17] — Hazard ratio: Arm C/Arm A
Statistical Analysis 2: Comparison: Arm A (Chemo + Placebo) vs Arm B (Chemo + Bevacizumab); Test type: Superiority; p = 0.92, Regression, Cox — Two-sided; based on stratified test using stratification factors at randomization; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.77 to 1.33] — Hazard ratio: Arm B/Arm A
Statistical Analysis 3: Comparison: Arm B (Chemo + Bevacizumab) vs Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy); Test type: Superiority; p = 0.36, Regression, Cox — Two-sided; based on stratified test using stratification factors at randomization; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.13] — Hazard ratio: Arm C/Arm B

3. Secondary Outcome: The Association Between IDFS and Genotype
Description: Invasive disease-free survival (IDFS) is defined as time from from date of randomization to first treatment failure (invasive ipsilateral, local/regional, or distant recurrence, invasive contralateral breast cancer, invasive non-breast second primary malignancy or death from any cause, whichever occurred first). Cases with incomplete follow-up, without documented IDFS event including those who developed squamous or basal cell skin cancers or insitu carcinomas of any site as their only event were censored at the date of last disease evaluation. Three-year IDFS rate was reported by genetic ancestry and IDFS was compared between patients with European ancestry and patients with African ancestry.
Time Frame: Assessed at 3 years
Population: Only patients with genetic ancestry as European ancestry or African ancestry were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- European Ancestry; African Ancestry: Genome-wide SNP arrays (either Illumina HumanOmni1-Quad or Human OmniExpress) were performed on germline DNA from whole blood to determine the genetic ancestry for the patients. The genetic ancestry is categorized into African ancestry (AA), European ancestry (EA) or other. Only African ancestry and European ancestry were included in these analyses.
Arm/Group | European Ancestry | African Ancestry
Number analyzed (Participants) | 2473 | 386
proportion of participants | 0.887 [0.875 to 0.900] | 0.832 [0.793 to 0.872]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed every cycle. Post protocol treatment, assessment and documentation of AEs continued 3 months post treatment for all AEs, and 6, 9, and 12 months post treatment for select AEs. The assessment and documentation of the select ≥ grade 4 hematologic and the select ≥ grade 2 non-hematologic AEs continued every 3 months until 1 year post protocol treatment. The assessment and documentation of ≥ grade 3 non-hematologic AEs took place 3 months post protocol treatment.
Description: Adverse event data collection in this trial was limited to ≥ grade 4 hematologic events, ≥ grade 2 non-hematologic events for a group of specific adverse events, and ≥ grade 3 non-hematologic events otherwise. All attributions were included. Detailed information on the select events could be found in the protocol.
Groups:
- Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm A and bevacizumab as in arm B. Treatment repeats every 2 or 3 weeks for 4 courses. Beginning 3 weeks later, patients then receive paclitaxel as in arm A and bevacizumab as in arm B. Treatment with paclitaxel and bevacizumab repeats every 3 weeks for 4 courses. Beginning 2 months later, patients then receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab alone repeats every 3 weeks for 10 courses. The monotherapy of bevacizumab is considered as Arm D in this study.
- Arm D (Bevacizumab Cycles 9-18 of Arm C): After completion of 4 cycles of paclitaxel and bevacizumab in arm C, patients then receive bevacizumab IV over 30-90 minutes on day 1 every 3 weeks for 10 courses. The monotherapy of bevacizumab is considered as Arm D in this study.
Arm/Group | Arm A (Chemo + Placebo) | Arm B (Chemo + Bevacizumab) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy) | Arm D (Bevacizumab Cycles 9-18 of Arm C)
Serious Adverse Events (participants affected / at risk) | 473/972 | 1090/1922 | 1136/1942 | 462/1168
Other Adverse Events (participants affected / at risk) | 245/972 | 513/1922 | 479/1942 | 233/1168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Chemo + Placebo) (N=972) | Arm B (Chemo + Bevacizumab) (N=1922) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy) (N=1942) | Arm D (Bevacizumab Cycles 9-18 of Arm C) (N=1168)
Allergic reaction (Immune system disorders) | 12 | 16 | 16 | 1
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hearing-other (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 15 | 32 | 26 | 5
Leukocytes decreased (Investigations) | 32 | 92 | 98 | 0
Lymphopenia (Investigations) | 7 | 13 | 8 | 0
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neutrophils decreased (Investigations) | 166 | 389 | 400 | 6
Platelets decreased (Investigations) | 4 | 11 | 19 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 5 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 2 | 4 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 3 | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 0 | 2 | 0
Vasovagal episode (Nervous system disorders) | 1 | 2 | 1 | 0
PVCs (Cardiac disorders) | 0 | 0 | 1 | 0
Torsade de pointes (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac-ischemia (Cardiac disorders) | 2 | 3 | 7 | 3
Cardiac troponin I (cTnI) increased (Investigations) | 0 | 1 | 5 | 0
Cardiac troponin T (cTnT) increased (Investigations) | 0 | 0 | 4 | 0
C-P arrest, non-fatal, cause unknown (Cardiac disorders) | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 20 | 147 | 138 | 131
Hypotension (Vascular disorders) | 3 | 11 | 8 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 4 | 9 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 9 | 38 | 43 | 34
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Cardiomyopathy, restrictive (Cardiac disorders) | 0 | 4 | 7 | 1
Cor Pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0
Valvular heart disease (Cardiac disorders) | 0 | 1 | 1 | 0
cardiac-other (Cardiac disorders) | 2 | 1 | 1 | 1
Fatigue (General disorders) | 66 | 188 | 195 | 31
Fever w/o neutropenia (General disorders) | 6 | 7 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 4 | 4 | 4
Obesity (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Rigors/chills (General disorders) | 1 | 2 | 1 | 0
Weight gain (Investigations) | 2 | 0 | 1 | 2
Weight loss (Investigations) | 2 | 7 | 4 | 10
Constitutional, other (General disorders) | 0 | 0 | 1 | 0
INR increased (Investigations) | 2 | 6 | 9 | 2
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 3 | 0
Coagulation-other (Investigations) | 0 | 1 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 6 | 12 | 11 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 | 32 | 26 | 17
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 12
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 8 | 26 | 20 | 0
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 4 | 17 | 12 | 17
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3
Death NOS (General disorders) | 0 | 2 | 2 | 1
Death - disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 2 | 3
Death - sudden death (General disorders) | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 4 | 9 | 6 | 4
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyopthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 8 | 26 | 29 | 4
Colitis (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 7 | 11 | 0
Dehydration (Metabolism and nutrition disorders) | 18 | 54 | 37 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Teeth (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 29 | 66 | 46 | 11
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 5 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Fistula, Abdomen NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fistula, Anus (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Fistula, Rectum (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Fistula, Small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 14 | 10 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 5 | 5 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Leak, incl. anastomotic, biliary tree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Leak, incl. anastomotic, Leak NOS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 3 | 4 | 0
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Muco/stomatitis by exam, rectum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 14 | 55 | 57 | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Muco/stomatitis (symptom) rectum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 25 | 54 | 57 | 5
Obstruction, cecum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstruction, colon (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstruction, small bowel NOS (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Perforation, appendix (Infections and infestations) | 1 | 0 | 0 | 0
Perforation, colon (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Perforation, small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stenosis (incl anastomotic) esophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Ulcer, anus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ulcer, duodenum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 15 | 49 | 44 | 8
GI-other (Gastrointestinal disorders) | 1 | 6 | 6 | 0
Hematoma (Vascular disorders) | 1 | 0 | 2 | 2
CNS, hemorrhage (Nervous system disorders) | 0 | 0 | 2 | 1
Abdomen, hemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 2 | 3 | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 2 | 6 | 6 | 2
Stomach, hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | 4 | 1
Bladder, hemorrhage (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 0 | 1 | 0
Uterus, hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Vagina, hemorrhage (Reproductive system and breast disorders) | 1 | 2 | 2 | 0
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6 | 2
Surgical hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 2 | 4
Liver dysfunction/failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hepatic-other (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 2 | 6 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 33 | 77 | 91 | 0
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, bladder (Infections and infestations) | 0 | 4 | 6 | 0
Infection w/ gr3-4 neut, bronchus (Infections and infestations) | 0 | 1 | 1 | 0
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 0 | 3 | 5 | 0
Infection w/ gr3-4 neut, colon (Infections and infestations) | 2 | 8 | 4 | 0
Infection w/ gr3-4 neut, dental-tooth (Infections and infestations) | 0 | 1 | 3 | 0
Infection w/ gr3-4 neut, external ear (Infections and infestations) | 1 | 0 | 0 | 0
Infection w/ gr3-4 neut, foreign body (Infections and infestations) | 2 | 1 | 1 | 0
Infection w/ gr3-4 neut, joint (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, kidney (Infections and infestations) | 0 | 2 | 1 | 0
Infection w/ gr3-4 neut, lip/perioral (Infections and infestations) | 0 | 0 | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 0 | 8 | 6 | 0
Infection w/ gr3-4 neut, lymphatic (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, mediastinum (Infections and infestations) | 0 | 0 | 1 | 0
Infection w/ gr3-4 neut, middle ear (Infections and infestations) | 0 | 0 | 1 | 0
Infection w/ gr3-4 neut, mucosa (Infections and infestations) | 0 | 1 | 2 | 0
Infection w/ gr3-4 neut, neck NOS (Infections and infestations) | 0 | 0 | 0 | 1
Infection w/ gr3-4 neut, oral cavity (Infections and infestations) | 0 | 0 | 1 | 0
Infection w/ gr3-4 neut, paranasal (Infections and infestations) | 0 | 1 | 1 | 0
Infection w/ gr3-4 neut, rectum (Infections and infestations) | 1 | 0 | 0 | 0
Infection w/ gr3-4 neut, sinus (Infections and infestations) | 0 | 3 | 3 | 0
Infection w/ gr3-4 neut, skin (Infections and infestations) | 5 | 12 | 8 | 0
Infection w/ gr3-4 neut, sm bowel NOS (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, soft tissue NOS (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 2 | 4 | 2 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 10 | 8 | 0
Infection w/ gr3-4 neut, vagina (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, vulva (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, wound (Infections and infestations) | 0 | 5 | 7 | 0
Infection Gr0-2 neut, abdomen (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, anal/perianl (Infections and infestations) | 0 | 6 | 2 | 0
Infection Gr0-2 neut, appendix (Infections and infestations) | 0 | 1 | 1 | 0
Infection Gr0-2 neut, bladder (Infections and infestations) | 1 | 3 | 5 | 0
Infection Gr0-2 neut, bone (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, bronchus (Infections and infestations) | 1 | 3 | 3 | 0
Infection Gr0-2 neut, catheter (Infections and infestations) | 4 | 9 | 16 | 1
Infection Gr0-2 neut, colon (Infections and infestations) | 1 | 6 | 4 | 0
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 2 | 0 | 1 | 0
Infection Gr0-2 neut, external ear (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 0 | 1 | 1 | 0
Infection Gr0-2 neut, foreign body (Infections and infestations) | 3 | 1 | 3 | 3
Infection Gr0-2 neut, gallbladder (Infections and infestations) | 0 | 1 | 1 | 0
Infection Gr0-2 neut, heart (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, kidney (Infections and infestations) | 2 | 0 | 1 | 0
Infection Gr0-2 neut, lip/perioral (Infections and infestations) | 0 | 0 | 2 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 9 | 19 | 27 | 3
Infection Gr0-2 neut, lymphatic (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, meninges (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, middle ear (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, muscle (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, nerve-periph (Infections and infestations) | 2 | 1 | 1 | 0
Infection Gr0-2 neut, nose (Infections and infestations) | 2 | 0 | 0 | 0
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 0 | 3 | 0 | 0
Infection Gr0-2 neut, pancreas (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, pelvis NOS (Infections and infestations) | 0 | 1 | 0 | 0
Infection Gr0-2 neut, pharynx (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, rectum (Infections and infestations) | 0 | 4 | 3 | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 0 | 4 | 5 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 19 | 25 | 22 | 9
Infection Gr0-2 neut, sm bowel (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, soft tissue (Infections and infestations) | 1 | 5 | 3 | 2
Infection Gr0-2 neut, stomach (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, ungual (Infections and infestations) | 1 | 3 | 5 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 2 | 4 | 5 | 0
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 2 | 7 | 4 | 3
Infection Gr0-2 neut, vagina (Infections and infestations) | 0 | 0 | 2 | 1
Infection Gr0-2 neut, vein (Infections and infestations) | 0 | 0 | 1 | 0
Infection Gr0-2 neut, vulva (Infections and infestations) | 0 | 0 | 3 | 0
Infection Gr0-2 neut, wound (Infections and infestations) | 6 | 15 | 12 | 4
Infection w/ unk ANC anal/perianal (Infections and infestations) | 0 | 0 | 1 | 0
Infection w/ unk ANC catheter related (Infections and infestations) | 0 | 0 | 3 | 1
Infection w/ unk ANC dental-tooth (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ unk ANC foreign body (Infections and infestations) | 0 | 5 | 0 | 1
Infection w/ unk ANC gallbladder (Infections and infestations) | 0 | 0 | 0 | 1
Infection w/ unk ANC lung (Infections and infestations) | 0 | 0 | 3 | 0
Infection w/ unk ANC meninges (Infections and infestations) | 0 | 0 | 0 | 1
Infection w/ unk ANC sinus (Infections and infestations) | 0 | 1 | 0 | 0
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 3 | 4 | 2
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 1 | 2 | 0 | 2
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 2 | 0 | 0
Infection w/ unk ANC wound (Infections and infestations) | 0 | 2 | 1 | 1
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 3 | 2 | 0 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 2 | 8 | 6 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 2 | 8 | 11 | 2
Infection-other (Infections and infestations) | 3 | 6 | 3 | 2
Edema head and neck (General disorders) | 0 | 2 | 1 | 0
Edema limb (General disorders) | 4 | 12 | 4 | 6
Edema trunk/genital (General disorders) | 0 | 1 | 0 | 2
Edema visceral (General disorders) | 0 | 1 | 1 | 0
Lymphedema-related fibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Lymphatics-other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercholesterolemia (Investigations) | 0 | 0 | 1 | 0
CPK increased (Investigations) | 0 | 0 | 2 | 0
Creatinine increased (Investigations) | 0 | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4 | 4 | 2
Proteinuria (Renal and urinary disorders) | 0 | 3 | 4 | 20
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 8 | 5 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 1 | 0
Extremity upper (function) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 5
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Local complication - device/prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3
Soft tissue necrosis, neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Soft tissue necrosis, thoracic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 2 | 4 | 1 | 3
CNS cerebrovascular ischemia (Nervous system disorders) | 2 | 4 | 5 | 5
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 1 | 1
Confusion (Psychiatric disorders) | 2 | 5 | 2 | 2
Dizziness (Nervous system disorders) | 11 | 15 | 18 | 3
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
Laryngeal nerve dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 1 | 0
Mental status (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 4 | 4 | 4
Depression (Psychiatric disorders) | 9 | 14 | 16 | 8
Neuropathy CN II vision (Eye disorders) | 0 | 0 | 1 | 0
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 7 | 10 | 10 | 2
Neuropathy-sensory (Nervous system disorders) | 82 | 153 | 172 | 49
Psychosis (Psychiatric disorders) | 0 | 4 | 0 | 0
Seizure (Nervous system disorders) | 1 | 2 | 3 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 2 | 2 | 0
Speech impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 12 | 34 | 22 | 8
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Neurologic-other (Nervous system disorders) | 0 | 1 | 4 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 2
Dry eye syndrome (Eye disorders) | 0 | 1 | 0 | 0
Double vision (Eye disorders) | 0 | 0 | 0 | 1
Vision-blurred (Eye disorders) | 2 | 1 | 2 | 1
Tearing (Eye disorders) | 0 | 1 | 0 | 0
Abdomen, pain (Gastrointestinal disorders) | 8 | 25 | 29 | 12
Anus, pain (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 9 | 8
Bladder, pain (Renal and urinary disorders) | 0 | 1 | 1 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 5 | 17 | 8 | 3
Breast, pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 1
Buttock, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cardiac/heart, pain (Cardiac disorders) | 1 | 2 | 5 | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 2
Chest/thoracic pain NOS (General disorders) | 10 | 25 | 25 | 9
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 0 | 5 | 2 | 0
External ear, pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4 | 3
Gallbladder, pain (Hepatobiliary disorders) | 0 | 1 | 2 | 0
Head/headache (Nervous system disorders) | 23 | 73 | 72 | 26
Joint, pain (Musculoskeletal and connective tissue disorders) | 26 | 37 | 43 | 40
Middle ear, pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 21 | 38 | 30 | 24
Neck, pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1
Neuropathic, pain (Nervous system disorders) | 2 | 2 | 0 | 2
Oral cavity, pain (Gastrointestinal disorders) | 1 | 5 | 2 | 0
Pain NOS (General disorders) | 0 | 2 | 1 | 1
Perineum, pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rectum, pain (Gastrointestinal disorders) | 1 | 8 | 4 | 0
Sinus, pain (Nervous system disorders) | 0 | 0 | 0 | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Stomach, pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Vagina, pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pain-other (General disorders) | 0 | 4 | 3 | 0
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
(DLCO) decreased (Investigations) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 18 | 19 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 | 60 | 63 | 18
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 9 | 3
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 | 27 | 16 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 8 | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4 | 3
Bladder spasms (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1 | 2 | 0
Obstruction-ureteral (Renal and urinary disorders) | 0 | 4 | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 1 | 3 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal/GU-other (Renal and urinary disorders) | 1 | 3 | 3 | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Intra-op injury Breast (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intra-op injury Parathyroid (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intra-op injury Pharynx (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 2 | 10 | 8 | 9
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0
Flu-like syndrome (General disorders) | 0 | 2 | 1 | 0
Syndromes-other (General disorders) | 0 | 0 | 1 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 6 | 13 | 10 | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 39 | 71 | 65 | 15
Vessel injury Extremity-upper (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular-Other (Specify) (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Chemo + Placebo) (N=972) | Arm B (Chemo + Bevacizumab) (N=1922) | Arm C (Chemo + Bevacizumab Then Bevacizumab Monotherapy) (N=1942) | Arm D (Bevacizumab Cycles 9-18 of Arm C) (N=1168)
Left ventricular systolic dysfunction (Cardiac disorders) | 37 | 103 | 87 | 64
Neuropathy-sensory (Nervous system disorders) | 188 | 356 | 334 | 182
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 52 | 117 | 119 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT00433511/Prot_SAP_000.pdf